CLINICAL TRIAL: NCT04579445
Title: Setting a Benchmark for Resource Utilization and Quality of Care in Patients Undergoing Transcatheter Aortic Valve Implantation in Europe - The BENCHMARK Registry
Brief Title: Setting a Benchmark for Resource Utilization and Quality of Care in Patients Undergoing TAVI in Europe
Acronym: BENCHMARK
Status: Completed | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: BENCHMARK Registry
Record Dates: First submitted 2020-09-28; First posted 2020-10-08 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Transcatheter Aortic Valve Implantation (TAVI)
Keywords: TAVI; Severe Aortic Stenosis; Optimizing TAVI patient outcomes; Optimizing TAVI care pathways
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TAVI patients: Consecutive, severe aortic stenosis patients undergoing transcatheter aortic valve implantation (TAVI) (there will be a retrospective part: documentation of 30 patients who underwent transfemoral TAVI; and a prospective part enrolling 50 patients undergoing transfemoral TAVI)
  Interventions: Other: Education on tailored Quality Improvement measures

INTERVENTIONS:
Other: Education on tailored Quality Improvement measures — Centers will undergo an education on defined Quality of Care measures, with the aim to implement a standardized pathway which is reproducible, scalable and which will allow increased access. The implementation of these measures will help to reduce resource requirements, intensive care bed occupancy and overall length of hospital stay with uncompromised patient safety.
  Other Names: Education on Quality of Care Improvement measures

SUMMARY:
Non-interventional, multi-center, international registry in patients with severe aortic stenosis (sAS) undergoing transcatheter aortic valve implantation (TAVI). The BENCHMARK Registry aims to implement standardized, reproducible and scalable quality improvement measures, which will help to reduce resource requirements, intensive care unit bed occupancy and overall length of hospitalization with uncompromised patient safety.

The registry will consist of the following phases:

* Retrospective phase (purpose: capture the status quo of each site prior to any Quality of Care improvement measures): The TAVI of patients being eligible for retrospective documentation must have been performed prior to the site's enrollment into the BENCHMARK prospective phase (follow-up: 30 days, 12 months).
* Education phase: Each center will undergo an online BENCHMARK education. The contents of the education will be: Reflection on treatment pathways with the TAVI team, education on 8 defined Quality of Care improvement measures, followed by a center self-assessment (to self-assess the current alignment of hospital performance with the BENCHMARK Quality od Care measures).
* Implementation phase: After having self-assessed the current alignment of hospital performance with the following BENCHMARK Quality of care measures, each center will start to introduce the tailored Quality of Care improvement measures to their hospital routine within a time frame of 2 months.
* Prospective phase (purpose: to document the effects of defined quality of care improvement measure and to make sure patient safety is as least as good as in the retrospective phase. (8 months of recruitment, Follow-up: 30 days, 12 months)

DETAILED DESCRIPTION:
Transcatheter aortic valve implantation (TAVI) has become standard of care in patients suffering from severe, symptomatic aortic stenosis, irrespective of risk. However, despite the advances in valve technology and implantation techniques, there is still no consensus on how to effectively screen, manage and discharge patients undergoing such an intervention.

In an effort not to lose grounds because of an increasing inner-hospital competition for resources including intensive care unit (ICU) and general hospital beds, there is a need for a streamlined Quality of Care (QoC) pathway that delivers the procedure more efficient, but with at least the same patient safety. In this context, the recent FAST-TAVI (Feasibility And Safety of early discharge after Transfemoral TAVI) and North American Multidisciplinary, Multimodality, But Minimalist (3M) studies have shown that optimized risk assessment and patient management results in a more effective, as least as safe treatment pathway and a reduced length of stay (LoS).

The results gain importance especially in a situation where patients suffering from the coronavirus disease compete for hospital resources throughout Europe. Using a clear set of Quality of Care criteria, the BENCHMARK registry aims to document the progress that can be made if tailored Quality of Care improvement measures are initiated.

The hypothesis is that the implementation of standardized, reproducible and scalable Quality of Care improvement measures will help reducing resource requirements, intensive care unit bed occupancy and overall length of hospitalization with uncompromised patient safety.

There will be up to 30 centers participating across Europe (Germany, Austria, Italy, France, Spain, Czech Republic, Romania). Each center will enroll 80 patients (retrospective documentation of 30 patients, prospective enrollment of 50 patients), resulting in 2400 patients in total.

ELIGIBILITY:
Inclusion Criteria:

Retrospective phase:

* Consecutive, severe symptomatic aortic stenosis patients who underwent transcatheter aortic valve implantation with a balloon-expandable transcatheter aortic valve prior to the center education on BENCHMARK QoC (Quality of Care) improvement measure (prior to the first education call)).
* Patient is or was scheduled to undergo a 30 Day and 12 Months follow-up (30 Day and 12 Months follow-up: hospital visit or phone call)
* All patients irrespective of valve type or access route will be documented in an electronic Case Report Form (eCRF) based patient logbook.

Prospective phase:

* Consecutive patients with a diagnosis of severe symptomatic aortic stenosis admitted for TAVI with a balloon-expandable transcatheter heart valve after center education on BENCHMARK Quality of Care measures and after the center has passed the implementation phase.
* All patients irrespective of valve type or access route will be documented in an eCRF based patient logbook.

Exclusion Criteria:

Retrospective phase:

* Patients with largely incomplete data with respect to the aims of the project.
* Patients without signed informed consent / data protection statement (according to requirements of local ethical committee).
* Pregnant women at the time of the TAVI.

Prospective phase:

* Patients without signed informed consent prior to the TAVI procedure (data protection statement included; ideally covered by hospital routine to enable consecutiveness).
* Pregnant women at the time of the TAVI.

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective phase:
  50 severe Aortic stenosis patients undergoing transcatheter aortic valve implantation will be recruited within the prospective part per center.
  Retrospective phase:
  Retrospective documentation of 30 severe aortic stenosis pateints per center, who underwent a transcatheter aortic valve implantation will be performed.
Sampling Method: Non-Probability Sample
Enrollment: 2408 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of differences in length of stay (LoS) | 12 months
  LoS in days
Complication rate (AEs), TAVI related safety outcomes | 30 days
  According to Valve Academic Research Consortium-2 consensus (VARC-2) criteria
Complication rate (AEs), TAVI related safety outcomes | 12 months
  According to Valve Academic Research Consortium-2 consensus (VARC-2) criteria
Quality of Life assessment: Toronto Aortic Stenosis Quality of Life Questionnaire | 30 days
  Assess the Quality of Life by using the Toronto Aortic Stenosis Quality of Life Questionnaire (TASQ). Each question has a maximum score of 7 (response options from "not very much" to "very much"), giving the complete questionnaire a maximum total score of 112 with a higher score indicating improved Quality of Life.
Quality of Life assessment: Toronto Aortic Stenosis Quality of Life Questionnaire | 12 months
  Assess the Quality of Life by using the Toronto Aortic Stenosis Quality of Life Questionnaire (TASQ). Each question has a maximum score of 7 (response options from "not very much" to "very much"), giving the complete questionnaire a maximum total score of 112 with a higher score indicating improved Quality of Life.
Resource utilization - Early discharge information | 12 months
  To determine the proportion of early discharges in sAS patients undergoing TAVI
Resource utilization - Working hours per patient | 12 months
  To determine the working hours per patient
Resource utilization - Number of TAVI patients in each center | 12 months
  To determine the number of patients undergoing TAVI (per center)
Physician and patient satisfaction | 30 days
  Satisfaction score, scoring from 0 (extremely dissatisfied) to 40 (extremely satisfied)
Physician and patient satisfaction | 12 months
  Satisfaction score, scoring from 0 (extremely dissatisfied) to 40 (extremely satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Derk Frank, Prof., Principal Investigator — UKSH Kiel; Gemma McCalmont, Principal Investigator — James Cook Hospital, Middlesbrough, United Kingdom
Locations (28):
- Austria (2):
  - St. Pölten University Hospital, Sankt Pölten
  - KH Nord, Klinik Floridsdorf, Vienna
- IKEM Prague, Prague, Czechia
- France (9):
  - Centre Hospitalier Universitaire de Besancon, Besançon
  - Polyclinique Du Bois, Lille
  - Infirmerie Protestante de Lyon, Lyon
  - Hopital Saint Joseph, Marseille
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - IMM (Institut Mutualiste Montsouris) Paris, Paris
  - Pitie Salpetriere Hospital Paris, Paris
  - CHU Rennes, Rennes
  - CHRU Tours, Tours
- Germany (6):
  - Herzzentrum Köln, Cologne
  - University Medical Center Göttingen, Göttingen
  - University Hospital Heidelberg, Heidelberg
  - Saarland University Medical Center, Homburg
  - CKMS Munich, Artemed Clinics, Munich
  - Brüderkrankenhaus Trier, Trier
- Italy (4):
  - L'Ospedale S.Giuseppe Moscati di Avellino, Avellino
  - Careggi Hospital, Florence
  - Centro Cardiologico, Monzino Hospital, Milan
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino
- Institutul de Urgenta pentru Boli Cardiolvasculaire, Bucharest, Romania
- Spain (5):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Bellvitge, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitari Son Espases, Palma de Mallorca

IPD SHARING:
Plan to Share IPD: No
no individual participant data (IPD) will be shared

REFERENCES:
- [Background] McCalmont G, Durand E, Lauck S, Muir DF, Spence MS, Vasa-Nicotera M, Wood D, Saia F, Chatel N, Luske CM, Kurucova J, Bramlage P, Frank D. Setting a benchmark for resource utilization and quality of care in patients undergoing transcatheter aortic valve implantation in Europe-Rationale and design of the international BENCHMARK registry. Clin Cardiol. 2021 Oct;44(10):1344-1353. doi: 10.1002/clc.23711. Epub 2021 Sep 9. PMID 34499383
- [Result] Frank D, Durand E, Lauck S, Muir DF, Spence M, Vasa-Nicotera M, Wood D, Saia F, Urbano-Carrillo CA, Bouchayer D, Iliescu VA, Saint Etienne C, Leclercq F, Auffret V, Asmarats L, Di Mario C, Veugeois A, Maly J, Schober A, Nombela-Franco L, Werner N, Gomez-Hospital JA, Mascherbauer J, Musumeci G, Meneveau N, Meurice T, Mahfoud F, De Marco F, Seidler T, Leuschner F, Joly P, Collet JP, Vogt F, Di Lorenzo E, Kuhn E, Disdier VP, Hachaturyan V, Luske CM, Rakova R, Wesselink W, Kurucova J, Bramlage P, McCalmont G; BENCHMARK Investigator Group. A streamlined pathway for transcatheter aortic valve implantation: the BENCHMARK study. Eur Heart J. 2024 Jun 1;45(21):1904-1916. doi: 10.1093/eurheartj/ehae147. PMID 38554125
- [Derived] Saia F, Lauck S, Durand E, Muir DF, Spence M, Vasa-Nicotera M, Wood D, Urbano-Carrillo CA, Bouchayer D, Iliescu VA, Etienne CS, Leclercq F, Auffret V, Asmarats L, Di Mario C, Veugeois A, Maly J, Schober A, Nombela-Franco L, Werner N, Gomez-Hospital JA, Mascherbauer J, Musumeci G, Meneveau N, Meurice T, Mahfoud F, De Marco F, Seidler T, Leuschner F, Joly P, Collet JP, Vogt F, Di Lorenzo E, Kuhn E, Disdier VP, McCalmont G, Rakova R, Wesselink W, Kurucova J, Hachaturyan V, Luske CM, Bramlage P, Frank D; BENCHMARK Investigator Group. The implementation of a streamlined TAVI patient pathway across five European countries: BENCHMARK registry. Clin Res Cardiol. 2025 Apr 22. doi: 10.1007/s00392-025-02638-z. Online ahead of print. PMID 40261426
- See also: Registry webpage — https://benchmark-registry.com